# USEFULNESS OF MULTIMODAL INTRAOPERTIVE NEUROPHYSIOLOGIC MONITORING DURING DIFFERENT NEUROSURGICAL OPERATIONS

**NCT** number: not available

**Document Date: 18 November 2021** 

## Informed Consent Form for Participation in a Research Study

**Title of the Study**: Usefulness of Multimodal Intraoperative Neurophysiologic Monitoring During Neurosurgical Operations

# **Principal Investigator:**

Dr. Ahmed Mosaad Mohamed Arafa Elsakka Ass.Lecturer Faculty of Medicine, Alexandria University

#### Introduction

You are being asked to participate in a research study. This document provides information about the study and explains what your participation would involve. Please read it carefully and feel free to ask any questions before agreeing to participate.

## **Purpose of the Study**

The purpose of this study is to evaluate the effectiveness of multimodal intraoperative neurophysiologic monitoring (MIONM) in preventing neurological deficits during brain and spine surgeries.

#### **Procedures**

If you agree to participate, the following will apply:

- Your surgery will be monitored using MIONM, which includes techniques such as Somatosensory Evoked Potentials (SSEP), Motor Evoked Potentials (MEP), and Electromyography (EMG).
- These techniques involve placing electrodes on your scalp, limbs, and/or other areas to monitor the function of your nervous system during the operation.
- Data collected during the surgery will be analyzed to assess the safety and effectiveness of MIONM.

#### **Risks and Discomforts**

- The procedures for MIONM are non-invasive and typically pose minimal risk. However, you may experience minor skin irritation at the electrode sites.
- There is a rare chance of mild discomfort during nerve stimulation, which will be minimized by the surgical and monitoring teams.

### **Benefits**

- Participating in this study may help prevent potential neurological deficits during your surgery.
- This study will contribute to improving surgical monitoring techniques and patient outcomes in similar cases.

# Confidentiality

- All personal and medical information will be kept confidential and stored securely.
- Data collected during the study will be anonymized to ensure your privacy.
- Only authorized personnel will have access to your information.

# **Voluntary Participation**

- Your participation is entirely voluntary.
- You may withdraw from studying at any time without affecting your medical care.

## Compensation

• There will be no financial compensation for participating in this study.

#### **Contact Information**

If you have questions or concerns about the study, you can contact:

 Dr. Ahmed Mosaad Mohamed Arafa Elsakka Email: [a\_sakka2008@alexmed.edue.g]

If you have questions about your rights as a participant, you may contact the ethics committee at Alexandria University.

#### Consent

| I have read and understood the information provided in this form. I have had the opportunity to a | sk |
|---|---|
| questions and agree to participate in this study. | |

| Participant Name: |
|------------------------|
| Participant Signature: |
| Date: |

| Witness Name: | <br>_ |
|-------------------------|-------|
| Witness Signature: | |
| Date: | |
| Investigator Name: | |
| Investigator Signature: | |
| Date: | |